CLINICAL TRIAL: NCT05065515
Title: Establishment of Individualized Immunotherapy Strategy and Platform for Upper Gastrointestinal Cancer Based on Changes of Intestinal Microbiota
Brief Title: Establishment of Individualized Immunotherapy Strategy and Platform Based on Changes of Intestinal Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20212109-C-1
Record Dates: First submitted 2021-09-16; First posted 2021-10-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-09

CONDITIONS: Gut Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — treatment and control groups' feces and a small amount of blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore and analyze the relationship between intestinal flora changes and the efficacy of individualized immunotherapy in patients with upper gastrointestinal cancer, and to find new biomarkers to predict the efficacy of immunotherapy, bringing new breakthroughs in tumor diagnosis and treatment.

DETAILED DESCRIPTION:
1. Compare the composition of intestinal flora of patients before and after immunotherapy and in patients with different therapeutic effects of immunotherapy.
2. Combine the results above with the patient's blood sample, which is carried out from the metabolic level.
3. Combine the pathological data of the patient to determine the staging and pathological types, and use blood samples to detect metabolites to find out different metabolites.
4. the metabolic data and the flora data are associated with the analysis to find the bacteria species with higher correlation with the differential metabolites to guide the subsequent animal experiments.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, no gender limit;
2. BMI index 18.5-23.9kg/m2;
3. Patients with esophageal squamous cell carcinoma, gastric adenocarcinoma or gastrointestinal stromal tumor diagnosed by pathology;
4. Patients who intend to undergo individualized immunotherapy, who have not undergone surgery in the past;
5. Patients with advanced or unresectable upper gastrointestinal tumors according to clinical stage;
6. ECOG score: 0-1 points;
7. Estimated survival period ≥ 3 months;
8. All patients should have measurable or evaluable target lesions;
9. Able to eat a liquid diet or above; no complete obstruction or perforation of the digestive tract; no distant metastasis;
10. The main organs are functioning normally, that is, they meet the following standards:

(1) Routine blood examination standards must meet (no blood transfusion and blood products within 14 days, no correction with G-CSF and other hematopoietic stimulating factors):

1. HB≥80 g/L;
2. ANC≥1.5×109/L;
3. PLT≥100×109/L; (2) The biochemical inspection shall meet the following standards:

a) TBIL<1.5×ULN; b) ALT and AST<2.0×ULN; c) Serum Cr≤1.5×ULN or endogenous creatinine clearance> 50 mL/min (Cockcroft-Gault formula); (3) Pulmonary function assessment: Pulmonary function is normal or mild to moderately abnormal (VC%>60%, FEV1>1.2L, FEV1%>40%, DLco>40%); (4) Cardiovascular function assessment: cardiac function grade Ⅰ～Ⅱ; 11. Have a certain degree of self-care ability and language comprehension ability;

Exclusion Criteria:

1. Patients with pathological types and primary foci that do not meet the inclusion criteria;
2. People who are known to be allergic to macromolecular protein preparations, or to immunological preparations and contrast agents and their preparation components;
3. Risk of digestive tract perforation;
4. Evidence of distant organ metastasis;
5. Surgical treatment (except biopsy), radiotherapy, chemotherapy, and molecular targeted therapy have been performed;
6. Have suffered from other malignant tumors;
7. History of serious lung or heart disease;
8. Have active infection or have fever of unknown cause > 38.5℃ within 2 weeks prior to randomization (according to the judgment of the investigator, the subjects' fever due to tumor can be included in the study);
9. Significant active infection is known, or significant blood, renal, metabolic, gastrointestinal, or endocrine dysfunction is determined by the investigator;
10. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency disease, or a history of organ transplantation;
11. The subject has active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody and hcV-RNA higher than the detection limit of analysis method);
12. Those who received live vaccine within 3 months prior to treatment;
13. Patients with acute or chronic tuberculosis infection (positive t-spot test, suspicious tuberculosis foci on chest X-ray);
14. History of drug, drug or alcohol abuse (drinking ≥5 times a week, ≥2 liang of liquor each time, etc.);
15. The patient participated in clinical trials of other antineoplastic agents within 4 weeks;
16. No intravenous infusion;
17. Severe diarrhea in the past 2 months (≥3 watery stools per day for ≥3 days);
18. Severe constipation in the past 2 months (defecation ≤2 times per week, with difficulty defecating);
19. Used antibiotics for 3 days or more in the past 2 months;
20. Used proton pump stomach drugs, acid suppressants, mucosal protectants, opioid psychotropic drugs, hormones, immunosuppressants, cytotoxic drugs and other drugs within the past 2 months for 3 days or more;
21. Used probiotics, prebiotics or biosaccharides for 3 days or more in the past 2 months;
22. Abnormal thyroid function caused by cholecystitis, gastrointestinal ulcer, urinary tract infection, acute pyelonephritis, cystitis, hyperthyroidism and other diseases within the past 1 month;
23. Medical procedures such as gastrointestinal surgery, appendicitis surgery or enema or bowel cleansing have been performed within the past 1 year;
24. Lactose intolerance during pregnancy and lactation (female);
25. Patients with hypertension who cannot be reduced to the normal range by antihypertensive medication (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg);A history of unstable angina pectoris;Patients who were newly diagnosed with angina pectoris within 3 months before screening or had myocardial infarction within 6 months before screening;Arrhythmias (including QTcF: ≥450 ms for men and ≥470 ms for women) requiring long-term use of antiarrhythmic drugs and New York Heart Association classification ≥II cardiac insufficiency;
26. In the investigator's judgment, the subject has other factors that may cause him/her to be forced to terminate the study, such as other serious diseases (including mental illness) requiring combined treatment, seriously abnormal laboratory test values, family or social factors that may affect the subject's safety or the collection of test data;
27. The investigator determines other conditions that may affect the conduct of the clinical study and the determination of the study results;
28. Partners or first-degree relatives of research centre staff, researchers;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age: 18-80 years old, no gender limit;
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Degree of tumor regression | 6 months
  We used the RECIST 1.1 evaluation criteria to evaluate the response to the immune therapy and accordingly divided patients into two groups，Response and No Response.

SECONDARY OUTCOMES:
The relative abundance of species | 6 months
  Use polymerase chain reaction (PCR) to specifically expand Increase the V3-V4 variable region of 16SrRNA and perform community analysis

OTHER OUTCOMES:
Species richness | 6 months
  Use polymerase chain reaction (PCR) to specifically expand Increase the V3-V4 variable region of 16SrRNA and perform community analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Yang, Dr, Principal Investigator — Xijing Hospital
Locations (1):
- Jianjun Yang, Xi'an, China